CLINICAL TRIAL: NCT04539249
Title: Single-centre, Randomized, Clinical Trial of Opioid-free Analgesia Versus Routine Opioid-based Analgesia Regimen for the Management of Acute Post-operative Pain Following Caesarean Section
Brief Title: Opioid-free Analgesia for the Management of Acute Post-operative Pain Following Caesarean Section
Acronym: OFAAPPCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olakunle Ifeoluwa Makinde (Other Government)
Responsible Party: Sponsor-Investigator, Olakunle Ifeoluwa Makinde, Senior Registrar, Federal Medical Centre, Yenagoa
Organization: Federal Medical Centre, Yenagoa (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMCY/O&G/OFAAPPCS/2020
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-08

CONDITIONS: Acute Post-operative Pain Following Caesarean Section
MeSH Terms: interventions — Magnesium Sulfate; Pentazocine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium sulphate (Experimental): Combination of intravenous magnesium sulphate, intravenous paracetamol and rectal diclofenac
  Interventions: Drug: Magnesium sulphate
- Pentazocine (Active Comparator): Combination of intramuscular pentazocine, intravenous paracetamol and rectal diclofenac
  Interventions: Drug: Pentazocine

INTERVENTIONS:
Drug: Magnesium sulphate — 1g of paracetamol as an I.V infusion and 4g of magnesium sulphate as an I.V. bolus preoperatively. Continuous infusion of 1g/hr of magnesium sulphate intraoperatively and for the first 2 hours post-operatively. Further post-operatively, 100 mg of suppository diclofenac 12 hourly, intravenous paracetamol 1g 6 hourly, both over 24 hours.
  N.B: Intramuscular pentazocine 30 mg (45 mg if patient is > 70 kg) will be used as rescue analgesia as needed (that is, only on patients' request for further analgesia or following an assessment of moderate to severe pain despite the planned analgesic regimen) at least 4 hourly during the first 24 hours after caesarean section.
  Other Names: MgSO4
  Arms: Magnesium sulphate
Drug: Pentazocine — Post-operatively, suppository diclofenac 100mg 12 hourly, intramuscular pentazocine 30 mg (45 mg if patient is > 70 kg) 6 hourly, intravenous paracetamol 1g 6 hourly, all for 24 hours.
  N.B: Intramuscular pentazocine 30 mg (45 mg if patient is > 70 kg) will be used as rescue analgesia as needed (that is, only on patients' request for further analgesia or following an assessment of moderate to severe pain despite the planned analgesic regimen) at least 4 hourly during the first 24 hours after caesarean section.
  Arms: Pentazocine

SUMMARY:
Background: Multimodal analgesia; a combination of opioid and non-opioid analgesics, for management of acute post-operative pain significantly reduces the incidence of adverse effects associated with liberal post-operative opioid use including sedation, respiratory depression, constipation, ileus, urinary retention, delayed recovery, addiction etc. However, opioid addiction remains a worsening public health problem and have followed administration of opioid analgesics for post-operative pain and subsequent chronic use in many addicts; especially the opioid naive. Caesarean section is a commonly performed surgery and is a common source of first exposure to opioids in women. Trend in post-operative analgesia is moving towards opioid-free (multimodal) analgesia; a combination of non-opioid and adjuvant analgesics. Magnesium sulphate is an adjuvant analgesic. When administered peri-operatively, it has been reported to prolong the duration of spinal anaesthesia, decrease post-operative pain and opioid use without adverse effect.

Aim: To determine the effectiveness and safety of a combination of peri-operative intravenous magnesium sulphate, intravenous paracetamol, and post-operative rectal diclofenac as opioid-free, multimodal analgesia for management of acute post-operative pain after a caesarean section.

Null Hypothesis: Combination of intravenous magnesium sulphate, intravenous paracetamol, and rectal diclofenac as analgesia regimen for acute post-operative pain after a caesarean section is not as effective and safe as a routine opioid-based multimodal analgesia regimen used in the study setting.

Alternate Hypothesis: Combination of intravenous magnesium sulphate, intravenous paracetamol, and rectal diclofenac as analgesia regimen for acute post-operative pain after a caesarean section is as effective and safe as a routine opioid-based multimodal analgesia regimen used in the study setting.

Materials and Methods: A randomized clinical trial, comparing a combination of peri-operative intravenous magnesium sulphate, intravenous paracetamol, and post-operative rectal diclofenac with an opioid-based multimodal regimen as control. Eligible patients will be consecutively selected from among women booked for caesarean section at the Federal Medical Centre, Yenagoa. Control group will receive a combination of post-operative intramuscular pentazocine, intravenous paracetamol and rectal diclofenac. Pain intensity will be determined in both groups and compared. Need for rescue opioid analgesic will be determined in both groups and compared. Incidence of any adverse event in both groups will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women booked for elective, scheduled and urgent caesarean section at the Federal Medical Centre, Yenagoa, Bayelsa State during the study period,
* Pregnant women who give consent to participate in the study.

Exclusion Criteria:

* Pregnant women with active peptic ulcer disease, active liver disease, hepatic failure, and renal failure,
* Pregnant women with previous history of ischaemic heart disease/myocardial infarction, heart failure, venous thrombosis and stroke,
* Hypersensitivity to pentazocine, paracetamol, diclofenac or magnesium sulphate,
* Pregnant women with history of non-medical use (abuse) of opioids,
* Pregnant women on magnesium sulphate or have a clinical indication to receive magnesium sulphate,
* Pregnant women booked for emergency caesarean section (because the urgency may not allow time for adequate patient counseling before recruitment)
* Pregnant women booked for caesarean section under general anaesthesia or epidural anaesthesia,
* Pregnant women who can neither communicate in english nor colloquial english.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 324 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olakunle I Makinde, MBChB, MWACS, Principal Investigator — Federal Medical Centre, Yenagoa
Locations (1):
- Federal Medical Centre, Yenagoa, Yenagoa, Bayelsa State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 3 months after publication
Access Criteria: Open access

REFERENCES:
- [Background] Vadivelu N, Mitra S, Schermer E, Kodumudi V, Kaye AD, Urman RD. Preventive analgesia for postoperative pain control: a broader concept. Local Reg Anesth. 2014 May 29;7:17-22. doi: 10.2147/LRA.S62160. eCollection 2014. PMID 24872720
- [Background] Kim M. An opioid success story: efforts to minimize painkillers after surgery appear to be working. Johannesburg, South Africa: The Conversation Africa, Inc.; 2019.
- [Background] Johnson SR. Hospitals look to cut opioids from surgery and beyond. Detroit, Michigan: Crain communications, Inc.; 2019.
- [Background] Dinis J, Soto E, Pedroza C, Chauhan SP, Blackwell S, Sibai B. Nonopioid versus opioid analgesia after hospital discharge following cesarean delivery: a randomized equivalence trial. Am J Obstet Gynecol. 2020 May;222(5):488.e1-488.e8. doi: 10.1016/j.ajog.2019.12.001. Epub 2019 Dec 6. PMID 31816306
- [Background] Kahraman F, Eroglu A. The effect of intravenous magnesium sulfate infusion on sensory spinal block and postoperative pain score in abdominal hysterectomy. Biomed Res Int. 2014;2014:236024. doi: 10.1155/2014/236024. Epub 2014 Mar 19. PMID 24772415
- [Background] McKeown A, Seppi V, Hodgson R. Intravenous Magnesium Sulphate for Analgesia after Caesarean Section: A Systematic Review. Anesthesiol Res Pract. 2017;2017:9186374. doi: 10.1155/2017/9186374. Epub 2017 Dec 3. PMID 29333156
- [Background] Shin HJ, Kim EY, Na HS, Kim TK, Kim MH, Do SH. Magnesium sulphate attenuates acute postoperative pain and increased pain intensity after surgical injury in staged bilateral total knee arthroplasty: a randomized, double-blinded, placebo-controlled trial. Br J Anaesth. 2016 Oct;117(4):497-503. doi: 10.1093/bja/aew227. Epub 2016 Oct 17. PMID 28077538
- [Background] Kalani N, Sanie MS, Zabetian H, Radmehr M, Sahraei R, Kargar Jahromi H, Zare Marzouni H. Comparison of the Analgesic Effect of Paracetamol and Magnesium Sulfate during Surgeries. World J Plast Surg. 2016 Sep;5(3):280-286. PMID 27853692
- [Background] Murphy JD, Paskaradevan J, Eisler LL, Ouanes JP, Tomas VA, Freck EA, Wu CL. Analgesic efficacy of continuous intravenous magnesium infusion as an adjuvant to morphine for postoperative analgesia: a systematic review and meta-analysis. Middle East J Anaesthesiol. 2013 Feb;22(1):11-20. PMID 23833845
- [Background] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Background] Hwang JY, Na HS, Jeon YT, Ro YJ, Kim CS, Do SH. I.V. infusion of magnesium sulphate during spinal anaesthesia improves postoperative analgesia. Br J Anaesth. 2010 Jan;104(1):89-93. doi: 10.1093/bja/aep334. PMID 19933175
- [Background] Apan A, Buyukkocak U, Ozcan S, Sari E, Basar H. Postoperative magnesium sulphate infusion reduces analgesic requirements in spinal anaesthesia. Eur J Anaesthesiol. 2004 Oct;21(10):766-9. doi: 10.1017/s026502150400002x. PMID 15678729
- [Background] Helmy N, Badawy AA, Hussein M, Reda H. Comparison of the preemptive analgesia of low dose ketamine versus magnesium sulphate on parturient undergoing caesarean section under general anaesthesia. Egypt. J. Anaesth. 2015;31(1):53-58.
- [Background] Paech MJ, Magann EF, Doherty DA, Verity LJ, Newnham JP. Does magnesium sulfate reduce the short- and long-term requirements for pain relief after caesarean delivery? A double-blind placebo-controlled trial. Am J Obstet Gynecol. 2006 Jun;194(6):1596-602; discussion 1602-3. doi: 10.1016/j.ajog.2006.01.009. Epub 2006 Apr 17. PMID 16615926

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 324 participants were enrolled and assessed for eligibility. A total of 224 of the enrolled participants were excluded from the study. Of the 224, one (1) declined to participate while the rest 223 did not meet the inclusion criteria.
Groups:
- Magnesium Sulphate: Combination of intravenous magnesium sulphate, intravenous paracetamol and rectal diclofenac
  Magnesium sulphate: 1g of paracetamol as an I.V infusion and 4g of magnesium sulphate as an I.V. bolus preoperatively. Continuous infusion of 1g/hr of magnesium sulphate intraoperatively and for the first 2 hours post-operatively. Further post-operatively, 100 mg of suppository diclofenac 12 hourly, intravenous paracetamol 1g 6 hourly, both over 24 hours.
  N.B: Intramuscular pentazocine 30 mg (45 mg if patient is > 70 kg) will be used as rescue analgesia as needed (that is, only on patients' request for further analgesia or following an assessment of moderate to severe pain despite the planned analgesic regimen) at least 4 hourly during the first 24 hours after caesarean section.
- Pentazocine: Combination of intramuscular pentazocine, intravenous paracetamol and rectal diclofenac
  Pentazocine: Post-operatively, suppository diclofenac 100mg 12 hourly, intramuscular pentazocine 30 mg (45 mg if patient is > 70 kg) 6 hourly, intravenous paracetamol 1g 6 hourly, all for 24 hours.
  N.B: Intramuscular pentazocine 30 mg (45 mg if patient is > 70 kg) will be used as rescue analgesia as needed (that is, only on patients' request for further analgesia or following an assessment of moderate to severe pain despite the planned analgesic regimen) at least 4 hourly during the first 24 hours after caesarean section.
Period: Overall Study
Arm/Group | Magnesium Sulphate | Pentazocine
Started (Randomized) | 50 | 50
Allocation (Received allocated intervention) | 50 | 50
Intervention Per Protocol (Received allocated intervention per protocol) | 49 | 50
Intervention NOT Per Protocol (Did not receive allocated intervention per protocol) | 1 | 0
Analyzed | 50 | 50
Excluded From Analysis | 0 | 0
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Sulphate | Pentazocine | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (3.4) | 30.8 (4.3) | 31.3 (3.9)
Age, Customized [Count of Participants; unit: Participants]
  20-24 | 0 | 1 | 1
  25-29 | 12 | 19 | 31
  30-34 | 25 | 16 | 41
  35-39 | 13 | 14 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Igbo | 21 | 18 | 39
  Ijaw | 23 | 20 | 43
  Others | 6 | 12 | 18
Region of Enrollment [Number; unit: participants]
  Nigeria | 50 | 50 | 100
Weight [Mean (Standard Deviation); unit: Kilograms] — Kilograms
  Kilograms | 84.5 (12.8) | 77.9 (8.9) | 81.2 (11.5)
Parity [Count of Participants; unit: Participants]
  Nulliparous (Never carried a pregnancy up to 28 weeks gestation or beyond) | 6 | 11 | 17
  Primiparous (Carried one (1) pregnancy up to 28 weeks and beyond, irrespective of outcome) | 11 | 6 | 17
  Multiparous (Carried two (2) or more pregnancies up to 28 weeks and beyond, irrespective of outcome) | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Scores Following Caesarean Section at 4 Hours Post-operative
Description: Post-operative pain scores following caesarean section at 4 hours post-operative using the Numerical Rating Scale for pain. The Numerical Rating Scale for pain has a minimum score of 0, a maximum score of 10 and a range of 0-10, where higher scores mean a worse outcome (0= No pain at all, 5= Moderate pain and 10= Worst pain imaginable)
Time Frame: 4 hours post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Magnesium Sulphate | Pentazocine
Number analyzed (Participants) | 50 | 50
score on a scale | 2.98 (1.18) | 3.16 (1.45)

2. Primary Outcome: Post-operative Pain Scores Following Caesarean Section at 8 Hours Post-operative
Description: Post-operative pain scores following caesarean section at 8 hours post-operative using the Numerical Rating Scale for pain. The Numerical Rating Scale for pain has a minimum score of 0, a maximum score of 10 and a range of 0-10, where higher scores mean a worse outcome (0= No pain at all, 5= Moderate pain and 10= Worst pain imaginable)
Time Frame: 8 hours post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Magnesium Sulphate | Pentazocine
Number analyzed (Participants) | 50 | 50
score on a scale | 2.58 (1.81) | 2.68 (1.63)

3. Primary Outcome: Post-operative Pain Scores Following Caesarean Section at 24 Hours Post-operative
Description: Post-operative pain scores following caesarean section at 24 hours post-operative using the Numerical Rating Scale for pain. The Numerical Rating Scale for pain has a minimum score of 0, a maximum score of 10 and a range of 0-10, where higher scores mean a worse outcome (0= No pain at all, 5= Moderate pain and 10= Worst pain imaginable)
Time Frame: 24 hours post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Magnesium Sulphate | Pentazocine
Number analyzed (Participants) | 50 | 50
score on a scale | 2.06 (1.42) | 2.37 (1.54)

4. Primary Outcome: Post-operative Pentazocine Use
Description: Whether or not Pentazocine was used post-operatively
Time Frame: 24 hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Sulphate | Pentazocine
Number analyzed (Participants) | 50 | 50
Participants
  Pentazocine used | 46 | 50
  Pentazocine NOT used | 4 | 0

5. Primary Outcome: Pentazocine Use as Rescue Analgesia
Description: Whether or not pentazocine was used as rescue analgesia
Time Frame: 24 hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Sulphate | Pentazocine
Number analyzed (Participants) | 50 | 50
Participants
  Pentazocine used as rescue analgesia | 46 | 0
  Pentazocine NOT used as rescue analgesia | 4 | 50

6. Primary Outcome: Frequency and Nature of Pentazocine Use
Description: Frequency of Pentazocine use per participant in each arm of the study and whether it was used as indicated in the protocol and/or for rescue analgesia
Time Frame: 24 hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Sulphate | Pentazocine
Number analyzed (Participants) | 50 | 50
Participants
  More than 4 times (per protocol + as rescue analgesia) | 0 | 0
  Four times (per protocol) | 0 | 50
  Four times (as rescue analgesia) | 0 | 0
  Three times (as rescue analgesia) | 0 | 0
  Two times (as rescue analgesia) | 11 | 0
  Once (as rescue analgesia) | 35 | 0
  Not used at all | 4 | 0

7. Primary Outcome: Mean Dose of Pentazocine Used
Description: Mean dose of Pentazocine used in each arm of the study
Time Frame: 24 hours post-operative
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Magnesium Sulphate | Pentazocine
Number analyzed (Participants) | 50 | 50
Milligrams | 52.83 (21.85) | 164.40 (28.59)

8. Secondary Outcome: Number of Participants With Peri-operative Adverse Events
Description: Number of participants with peri-operative adverse events including hypersensitivity reaction, respiratory depression, bradycardia, hypotension, nausea and vomiting, lightheadedness, presyncope, and any other adverse event recorded from the time of first administration of peri-operative analgesia to 2 hours postoperative
Time Frame: Time of first administration of peri-operative analgesia to 2 hours postoperative
Population: Number analyzed under severe (symptomatic) systolic hypotension (n=14; MgSo4 arm, n=5; Pentazocine arm ) and under severe (symptomatic) diastolic hypotension (n=24; MgSo4 arm, n=18; Pentazocine arm ) are subsets of the outcome measures systolic hypotension and diastolic hypotension with participant counts of (n=14; MgSo4 arm, n=5; Pentazocine arm ) and (n=24; MgSo4 arm, n=18; Pentazocine arm ) respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Sulphate | Pentazocine
Number analyzed (Participants) | 50 | 50
Participants
  Bradycardia: Present | 0 | 2
  Bradycardia: Absent | 50 | 48
  Systolic hypotension: Present | 14 | 5
  Systolic hypotension: Absent | 36 | 45
  Severe (Symptomatic) systolic hypotension: number analyzed (Participants) | 14 | 5
  Severe (Symptomatic) systolic hypotension: Present | 1 | 0
  Severe (Symptomatic) systolic hypotension: Absent | 13 | 5
  Diastolic hypotension: Present | 24 | 18
  Diastolic hypotension: Absent | 26 | 32
  Severe (Symptomatic) diastolic hypotension: number analyzed (Participants) | 24 | 18
  Severe (Symptomatic) diastolic hypotension: Present | 1 | 0
  Severe (Symptomatic) diastolic hypotension: Absent | 23 | 18
  Vomiting: Present | 1 | 0
  Vomiting: Absent | 49 | 50
  Lightheadedness: Present | 1 | 0
  Lightheadedness: Absent | 49 | 50
  Presyncope: Present | 1 | 0
  Presyncope: Absent | 49 | 50

9. Secondary Outcome: Number of Participants With Post-operative Adverse Events
Description: Number of participants with post-operative adverse events including respiratory depression constipation, ileus, pruritus, urinary retention and any other adverse event recorded during the first 24 hours post-operative.
Time Frame: First 24 hours post-operative
Measure: Count of Participants; unit: Participants
Groups:
- Magnesium Sulphate Only: Participants in the magnesium sulphate arm of the study who received a combination of peri-operative intravenous magnesium sulphate, intravenous paracetamol, and post-operative rectal diclofenac, but DID NOT receive post-operative intramuscular pentazocine as rescue analgesia
- Magnesium Sulphate and Pentazocine: Participants in the magnesium sulphate arm of the study who received a combination of peri-operative intravenous magnesium sulphate, intravenous paracetamol, and post-operative rectal diclofenac, and ALSO received post-operative intramuscular pentazocine as rescue analgesia
- Pentazocine Only: Participants in the pentazocine arm of the study who received a combination of post-operative intramuscular pentazocine, intravenous paracetamol and rectal diclofenac
Arm/Group | Magnesium Sulphate Only | Magnesium Sulphate and Pentazocine | Pentazocine Only
Number analyzed (Participants) | 4 | 46 | 50
Participants
  Present | 0 | 0 | 0
  Absent | 4 | 46 | 50

10. Secondary Outcome: Apgar Scores of the Neonates
Description: Apgar scores of the neonates delivered by the women who had caesarean section under the study, taken at first and fifth minutes after birth. Apgar score has a minimum score of 0, a maximum score of 10 and a range of 0-10, where higher scores mean a better outcome (0-3= low Apgar score, 4-6= moderately abnormal Apgar score and 7-10= reassuring Apgar score
Time Frame: At first and fifth minutes after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Sulphate | Pentazocine
Number analyzed (Participants) | 50 | 50
Participants
  Apgar score at the 1st minute: Less than 4 | 0 | 0
  Apgar score at the 1st minute: 4-6 | 2 | 6
  Apgar score at the 1st minute: 7-10 | 48 | 44
  Apgar score at the 5th minute: Less than 4 | 0 | 1
  Apgar score at the 5th minute: 4-6 | 0 | 0
  Apgar score at the 5th minute: 7-10 | 50 | 49

ADVERSE EVENTS:
Time Frame: Pre-operative, intra-operative and first 24 hours post-operative
Groups:
- Magnesium Sulphate Only: .Participants in the magnesium sulphate arm of the study who received a combination of peri-operative intravenous magnesium sulphate, intravenous paracetamol, and post-operative rectal diclofenac, but DID NOT receive post-operative intramuscular pentazocine as rescue analgesia
Arm/Group | Magnesium Sulphate Only | Magnesium Sulphate and Pentazocine | Pentazocine Only
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/46 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/46 | 0/50
Other Adverse Events (participants affected / at risk) | 4/4 | 19/46 | 20/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnesium Sulphate Only (N=4) | Magnesium Sulphate and Pentazocine (N=46) | Pentazocine Only (N=50)
Severe (symptomatic) hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnesium Sulphate Only (N=4) | Magnesium Sulphate and Pentazocine (N=46) | Pentazocine Only (N=50)
Mild (asymptomatic) systolic hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 5 (5)
Mild (asymptomatic) diastolic hypotension (Cardiac disorders) | 4 (4) | 19 (19) | 18 (18)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
1. The subjectivity of the perception, expression and assessment of pain was a limitation to this study. The intensity of pain cannot be perfectly compared between one person and the other, neither can it be objectively measured.
2. This study was done only among pregnant women undergoing a caesarean section at the Federal Medical Centre Yenagoa, Bayelsa State, which limits the generalizability of the findings to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT04539249/Prot_SAP_ICF_000.pdf